CLINICAL TRIAL: NCT06955000
Title: Efficacy of Interval Aerobic Training Versus Laser Puncture Therapy on the Severity of Restless Leg Syndrome in Chronic Obstructive Lung Disease Patients
Brief Title: Efficacy of Interval Aerobic Training Versus Laser Puncture Therapy on Restless Leg Syndrome in Copd Patient
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Ola Mohamed Elsayed Elgohary, lecturer at cardiovascular pulmonary and geratrics departement faculty of physical therapy pharos university, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: restless leg syndrome and copd
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: restless leg syndrom,lazer puncture therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic training (Experimental): 3 sessions per week,40 mints each session, mild to moderate intensity exercise
  Interventions: Device: traidmail
- laser puncture therapy (Experimental): There were three sessions per week, each lasting 40 minutes. Five minutes later, a laser probe was applied to the acupuncture sites on the leg.
  Interventions: Device: laser puncture therapy

INTERVENTIONS:
Device: traidmail — Patients in this group were instructed to sit on a stationary bicycle ergometer. The patients will be given explained the aerobic interval exercise training program and the intensity will be assessed using a modified Borg scale
  Arms: aerobic training
Device: laser puncture therapy — This group's patients were all exposed to LLLT utilising Phyaction CL Phyaction, Bilzen, Belgium, which had the following specs: frequency 500 Hz, output 5-20 MW, wavelength 905 nm. For five minutes, a laser probe was applied to acupuncture sites
  Other Names: laser puncture prob therapy
  Arms: laser puncture therapy

SUMMARY:
DETERMINE HOW TO IMPROVE THE QUALITY OF LIFE FOR PATIENTS WITH COPD BY DECREASING TINTENSITY OF THE RESTLESS SYNDROME

DETAILED DESCRIPTION:
Patients with restless legs syndrome can benefit greatly from aerobic exercise, and a novel treatment for enhancing quality of life is laser puncture therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men with COPD who were between the ages of 40 and 60 and had a BMI between 25.5 and 29.0 were eligible to enroll if they had received a diagnosis of COPD at least two years priorAn intense desire to move the legs is frequently accompanied by unpleasant and uncomfortable leg sensations. Patients usually experience worsening symptoms when they are at rest, sitting, or lying down. Walking and stretching are examples of physical activity that can help reduce these symptoms to some or all of their intensity

Exclusion Criteria:

* 1) Individuals suffering from acute infections and malignant diseases; 2) Individuals with a history of kidney disease, hiatus hernia, severe gastro-esophageal reflux, and osteoporosis 3) Patients with severe anemia and congestive heart failure 4) Individuals with severe neurological and musculoskeletal conditions.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2025-07-05 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Restless Legs Syndrome Rating Scale (IRLS): | 3 month
  Developed as a tool for assessing the severity Restless Legs Syndrome (RLS), the 10-item questionnaire asks respondents to use Likert-type ratings to indicate how acutely the disorder has affected them over the course of the past week. Questions can be divided into one of two catego- ries: disorder symptoms (nature, intensity, and frequency) and their impact (sleep issues, distur- bances in daily functioning, and resultant changes in mood)
Fatigue severity scale (FSS): | 3 month
  The FSS is a short questionnaire that requires you to rate your level of fatigue. The FSS questionnaire contains nine statements that rate the severity of your fatigue symptoms. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition during the past week and the extent to which you agree or disagree that the statement applies to you
Six mint walk test: | 3 month
  the 6-minute walk test (6MWT) is a key study providing a functional, therapeutic response, and prognostic data that is valuable in the care of patients with respiratory as well as cardiac diseases. It is used widely due to its simplicity and reproducibility,

SECONDARY OUTCOMES:
Hemoglobin Test: | 3 month
  Red blood cells contain hemoglobin, a protein that is rich in iron. It transports oxygen throughout the body from the lungs.

CONTACTS AND LOCATIONS:
Locations (1):
- Ola Mohamed Elsayed Elgohary, Alexandria, Egypt

REFERENCES:
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/35015445/ — Döner A, Taşci S, Bilgin A. The Effect of Massage, Acupressure and Reflexology on Restless Legs Syndrome Severity and Sleep Quality in Patients Receiving Haemodialysis Treatment: A Systematic Review and Meta-Analysis. Nursing Open. 2025 Feb;12(2):e70135. 26-Mitchell UH, Johnson AW, Myrer B. Comparison of two infrared devices in their effectiveness in reducing symptoms associated with RLS. Physiotherapy theory and practice. 2011 Jun 1;27(5):352-9. 27-Tang L, Zhao N, Gao X, Li J, Yu X, Liang R, Xie C, Li L, Wang Q, Yang W. Acupuncture treatment of restless legs syndrome: a randomized clinical controlled study protocol based on PET-CT and fMRI. Frontiers in Psychiatry. 2024 Dec 24; 15:1481167.